CLINICAL TRIAL: NCT03634423
Title: Enduring Exercise Habits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 827107
Record Dates: First submitted 2018-06-12; First posted 2018-08-16 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Healthy
Keywords: Interest in exercising more

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- Sweet Spot: Flexible high incentive condition (Experimental): Participants will receive 500 points if they make a gym visit within a pre-specified window of time and 490 points if they make a gym visit at any other time. 7000 points convert to $25
  Interventions: Behavioral: Sweet Spot: Flexible high incentive condition
- Sweet Spot: Flexible low incentive condition (Experimental): Participants will receive 300 points if they make a gym visit within a pre-specified window of time and 290 points if they make a gym visit at any other time. 7000 points convert to $25
  Interventions: Behavioral: Sweet Spot: Flexible low incentive condition
- Sweet Spot: Rigid high incentive condition (Experimental): Participants will receive 500 points if they make a gym visit within a pre-specified window of time and 250 points if they make a gym visit at any other time. 7000 points convert to $25
  Interventions: Behavioral: Sweet Spot: Rigid high incentive condition
- Sweet Spot: Rigid low incentive condition (Experimental): Participants will receive 300 points if they make a gym visit within a pre-specified window of time and 150 points if they make a gym visit at any other time. 7000 points convert to $25
  Interventions: Behavioral: Sweet Spot: Rigid low incentive condition
- FOTW: High incentive control condition (Experimental): Participants will receive 750 points if they make a gym visit within a pre-specified window of time and 250 points if they make a gym visit at any other time. 7000 points convert to $5
  Interventions: Behavioral: FOTW: High incentive control condition
- FOTW: Low incentive control condition (Experimental): Participants will receive 450 points if they make a gym visit within a pre-specified window of time and 150 points if they make a gym visit at any other time. 7000 points convert to $5
  Interventions: Behavioral: FOTW: Low incentive control condition
- FOTW: High incentive treatment condition (Experimental): Participants will receive 500 points if they make a gym visit within a pre-specified window of time and 250 points if they make a gym visit at any other time. Additionally, if a participant misses a scheduled gym visit, they will receive 750 points the next time they visit the gym within the pre-specified window. 7000 points convert to $5
  Interventions: Behavioral: FOTW: High incentive treatment condition
- FOTW: Low incentive treatment condition (Experimental): Participants will receive 300 points if they make a gym visit within a pre-specified window of time and 150 points if they make a gym visit at any other time. Additionally, if a participant misses a scheduled gym visit, they will receive 450 points the next time they visit the gym within the pre-specified window. 7000 points convert to $5
  Interventions: Behavioral: FOTW: Low incentive treatment condition
- Think Twice: Control condition (Experimental): Participants get 300 points per gym visit. 7000 points convert to $5
  Interventions: Behavioral: Think Twice: Control condition
- Think Twice: Treatment condition (Experimental): Participants get 300 points per gym visit and are taught about the planning fallacy. 7000 points convert to $5
  Interventions: Behavioral: Think Twice: Treatment condition
- WDR: Control condition (Experimental): Participants get 300 points per gym visit and are allowed to vary their gym schedules in different days. 7000 points convert to $5
  Interventions: Behavioral: WDR: Control condition
- WDR: Treatment condition (Experimental): Participants get 300 points per gym visit. Participants are required to select a single exercise time for the weekdays (Monday - Friday) and a single exercise time for the weekends (Saturday - Sunday). 7000 points convert to $5
  Interventions: Behavioral: WDR: Treatment condition

INTERVENTIONS:
Behavioral: Sweet Spot: Flexible high incentive condition — Participants receive text reminders 30 minutes before their workouts and weekly emails reminding them of their schedule.
  Arms: Sweet Spot: Flexible high incentive condition
Behavioral: Sweet Spot: Flexible low incentive condition — Participants receive text reminders 30 minutes before their workouts and weekly emails reminding them of their schedule.
  Arms: Sweet Spot: Flexible low incentive condition
Behavioral: Sweet Spot: Rigid high incentive condition — Participants receive text reminders 30 minutes before their workouts and weekly emails reminding them of their schedule.
  Arms: Sweet Spot: Rigid high incentive condition
Behavioral: Sweet Spot: Rigid low incentive condition — Participants receive text reminders 30 minutes before their workouts and weekly emails reminding them of their schedule.
  Arms: Sweet Spot: Rigid low incentive condition
Behavioral: FOTW: High incentive control condition — Participants receive text reminders 30 minutes before their workouts and weekly emails reminding them of their schedule.
  Arms: FOTW: High incentive control condition
Behavioral: FOTW: Low incentive control condition — Participants receive text reminders 30 minutes before their workouts and weekly emails reminding them of their schedule.
  Arms: FOTW: Low incentive control condition
Behavioral: FOTW: High incentive treatment condition — Participants receive text reminders 30 minutes before their workouts and weekly emails reminding them of their schedule.
  Arms: FOTW: High incentive treatment condition
Behavioral: FOTW: Low incentive treatment condition — Participants receive text reminders 30 minutes before their workouts and weekly emails reminding them of their schedule.
  Arms: FOTW: Low incentive treatment condition
Behavioral: Think Twice: Control condition — Participants receive text reminders 30 minutes before their workouts and weekly emails reminding them of their schedule.
  Arms: Think Twice: Control condition
Behavioral: Think Twice: Treatment condition — Participants receive text reminders 30 minutes before their workouts and weekly emails reminding them of their schedule.
  Arms: Think Twice: Treatment condition
Behavioral: WDR: Control condition — Participants receive text reminders 30 minutes before their workouts and weekly emails reminding them of their schedule.
  Arms: WDR: Control condition
Behavioral: WDR: Treatment condition — Participants receive text reminders 30 minutes before their workouts and weekly emails reminding them of their schedule.
  Arms: WDR: Treatment condition

SUMMARY:
The objective of this study is to test whether the interventions offering short-term incentives (points redeemable for prizes), specific cued plans, and science-backed tips can help with creating enduring exercise habits. There are four (4) sub-studies within this protocol.

DETAILED DESCRIPTION:
The four sub-studies are:

1. Sweet spot

   Past studies have shown that steady routines associated with stable cues are a hallmark of successful habits. However, recent research has demonstrated that incentivizing an overly rigid routine (e.g., every workout must be at the same time each day) creates a less lasting exercise habit than incentivizing a flexible exercise routine (e.g., workouts can be at any time of day). In this study, the investigators examine whether offering higher rewards for exercise that occurs at a planned, routine time than for exercise at other times, but still offering some rewards for exercise outside of these planned moments, may improve over total flexibility for producing lasting habits.
2. Falling off the Wagon (FOTW)

   In the long run, missing one workout won't make much difference to a person's overall health. Psychologically, however, missing a workout may lead people to feel they've already failed at meeting their fitness goals, zapping their motivation to exercise in the future. In this study, the investigators examine whether offering 50% larger incentive for exercise to people after they miss a planned workout leads to more sustained exercise habits than incentivizing all workouts equally.
3. Think Twice

   Studies have shown that people tend to fall into the planning fallacy -- optimistically overestimating their performance in some future activity. In this study, the investigators examine whether people who the investigators taught about the planning fallacy would make more realistic exercise plans and adhere to those plans better.
4. Weekly vs. Daily Routines (WDR)

This study will examine whether incentivizing people to create a daily routine that is consistent every day for a month or a weekly routine that is consistent every week for a month helps people build a more lasting exercise habit. In the daily routines condition, participants will be required to schedule workouts (and associated text reminders) at the same time of day on every weekday, and the same time of day on each weekend throughout our four week treatment period. In the weekly routines condition, participants will be allowed to schedule workouts (and associated text reminders) at different times on different days of the week, but their schedule must be the same for each of the four weeks of our four week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Has 24 Hour Fitness Membership

Exclusion Criteria:

-

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32000 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Each participant's number of gym visits per week | During the 4 intervention weeks
Each participant's number of gym visits per week | During the 4 weeks post-intervention
Each participant's number of gym visits per week | During the 10 weeks post-intervention
Each participant's number of gym visits per week | During the 52 weeks post-intervention
Binary variable capturing whether or not a participant had any gym visits in a given week | During the 4 intervention weeks
Binary variable capturing whether or not a participant had any gym visits in a given week | During the 4 weeks post-intervention
Binary variable capturing whether or not a participant had any gym visits in a given week | During the 10 weeks post-intervention
Binary variable capturing whether or not a participant had any gym visits in a given week | During the 52 weeks post-intervention
Each participant's number of gym visits per week at scheduled workout times | During the 4 intervention weeks
Each participant's number of gym visits per week at scheduled workout times | During the 4 weeks post-intervention
Each participant's number of gym visits per week at scheduled workout times | During the 10 weeks post-intervention
Each participant's number of gym visits per week at scheduled workout times | During the 52 weeks post-intervention
Binary variable capturing whether or not a participant had any gym visits in a given week at scheduled workout times | During the 4 intervention weeks
Binary variable capturing whether or not a participant had any gym visits in a given week at scheduled workout times | During the 4 weeks post-intervention
Binary variable capturing whether or not a participant had any gym visits in a given week at scheduled workout times | During the 10 weeks post-intervention
Binary variable capturing whether or not a participant had any gym visits in a given week at scheduled workout times | During the 52 weeks post-intervention
Each participant's number of gym visits per week outside of scheduled workout times | During the 4 intervention weeks
Each participant's number of gym visits per week outside of scheduled workout times | During the 4 weeks post-intervention
Each participant's number of gym visits per week outside of scheduled workout times | During the 10 weeks post-intervention
Each participant's number of gym visits per week outside of scheduled workout times | During the 52 weeks post-intervention
Binary variable capturing whether or not a participant had any gym visits in a given week outside of scheduled workout times | During the 4 intervention weeks
Binary variable capturing whether or not a participant had any gym visits in a given week outside of scheduled workout times | During the 4 weeks post-intervention
Binary variable capturing whether or not a participant had any gym visits in a given week outside of scheduled workout times | During the 10 weeks post-intervention
Binary variable capturing whether or not a participant had any gym visits in a given week outside of scheduled workout times | During the 52 weeks post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Katherine L. Milkman, PhD, Principal Investigator — University of Pennsylvania; John Beshears, PhD, Principal Investigator — Harvard University
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States